CLINICAL TRIAL: NCT06824935
Title: Investigation of Perioperative Anesthesia Requirements of Outpatient Cataract Patients Who Underwent Preoperative Anesthesia Evaluation.
Brief Title: Evaluation of Perioperative Anesthesia Requirements of Outpatient Cataract Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Naime Yalçın (Other)
Responsible Party: Sponsor-Investigator, Naime Yalçın, Specialist Anesthesiology and Reanimation, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Organization: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Other Study IDs: KAEK/2024.12.275
Record Dates: First submitted 2025-01-29; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Preoperative Evaluation; Outpatient; Cataract Surgery Anesthesia
MeSH Terms: interventions — Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Anesthesia — The study planned to investigate the anesthesia requirements and frequency and the risk factors that play a role in the anesthesia of patients who had completed preoperative anesthesia evaluation and were going to undergo outpatient cataract surgery.

SUMMARY:
According to the literature, preoperative evaluation has been shown in studies to be the first step in ensuring that patients' anesthesia care is carried out safely. In cataract surgery, which is a day anesthesia procedure frequently observed in the geriatric population, topical-local anesthesia is mostly applied. It is believed that preoperative anesthesia evaluation will be beneficial due to the complications that may develop during the procedure, patient safety and therefore the duration of postoperative hospital stay. The aim of the study is to evaluate patients who may need anesthesia intervention among patients whose preoperative anesthesia evaluations have been completed due to the possibility of consultation from the anesthesia department if necessary for patients who will undergo cataract surgery with local-topical anesthesia.

DETAILED DESCRIPTION:
Preoperative assessment is the first step in ensuring that patients receive safe anesthesia care. Over time, this process has changed significantly from an era when patients were admitted to the hospital the night before surgery to a time when the majority of patients, including those scheduled for major surgical procedures, arrive on the day of surgery. Outpatient preoperative assessment clinics are private and academic practices that require training in institutional staff; although common, the optimal model is unknown and may depend on the characteristics of the hospital, such as the specific types of care provided, geographic and socioeconomic differences in the population served by the hospital, patient expectations, and facility availability. The American Society of Anesthesiologists physical status (ASA-PS) classification provides a starting point for triage. Outpatient surgery may be safe even in patients with a high ASA-PS classification. A multicenter European study of 57,709 procedures including ASA PS III patients found that major complications such as stroke, myocardial infarction (MI), and pulmonary embolism were extremely rare and were not clearly associated with any deaths. Cataract surgery is the most frequently performed day surgery, with an estimated 3.3 million procedures performed annually by 2020 and 4.4 million by 2030. Almost all are performed in an outpatient setting with minimal intravenous sedation and different local anesthesia methods. The frequency of unplanned hospitalization on the day of surgery is estimated to be 0.05%. The majority of anesthesia interventions are related to the treatment of hypertension or bradycardia. Hypertension is often associated with anxiety and is often treated with sedation. Rarely, bradycardia requiring treatment typically occurs as a vagal response or following intravenous sedation. Considering the geriatric population and associated medical problems, monitored anesthesia care with anesthesia personnel may be considered more reliable in cataract surgery. Studies have reported that the rate of anesthesia call represents 3.4% of interventions, similar to those reported in the last 15 years, but some authors have reported higher anesthesia call rates of over 20%. In literature stated that the lack of premedication probably contributed to this increase, and that other factors such as the lack of anesthesia consultation, the level of information given to the patient, the definition of the criteria for calling the anesthesiologist, and the technique applied for topical anesthesia may have also affected the rates. The studies supported the need for anesthesia personnel to be present in the operating room to be evaluated by anesthesia personnel during cataract surgery by citing the study in 406 cases, in which the rate of anesthesia requirement during peribulbar anesthesia was shown as 28.5% and interventions were typically directed towards arrhythmia, agitation, or hypertension. The primary aim of this study was to evaluate patients who may need interventions in terms of anesthesia and reanimation among those who have completed preoperative anesthesia evaluations due to the possibility of consultation with the anesthesia department if needed in patients who will undergo cataract surgery under local-topical anesthesia. Investigator's secondary aim is to analyze the frequency of anesthesia interventions needed and the risk factors that play a role in these interventions by examining patient data, accompanied by patients' demographic data, medical history and preoperative anesthesia examinations.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old, ASA I-IV status, and undergoing cataract surgery under local-topical anesthesia

Exclusion Criteria:

* If the procedure is performed under general anesthesia or sedation, emergency surgery or ASA-E

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo local cataract surgery in the ophthalmology clinic by applying to our hospital's anesthesia polyclinic
Sampling Method: Non-Probability Sample
Enrollment: 470 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-05-02 (Estimated); Study Completion 2025-07-02 (Estimated)

PRIMARY OUTCOMES:
Number and nature of anesthesia requirements in local cataract surgery | Up to 8 weeks after registration
  Patients will be examined with parameters such as age, gender, weight and height will be combined to report BMI in kg/m^2, history of chronic disease, history of medication, smoking, alcohol, allergy, previous eye surgery, ASA, type of surgical anesthesia, reasons for anesthesia requirement, increasing oxygen flow rate, clarifying ECG, opening i.v. access, sedation, general anesthesia, additional medication, and length of hospital stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlık Bilimleri Üniversitesi Kanuni Sultan Süleyman Eğitim ve Araştırma Hastanesi, Istanbul, Turkey (Türkiye)